CLINICAL TRIAL: NCT02417792
Title: The Association Between Psoriasis and Intestinal Bacterial Population
Acronym: PIB
Status: Completed | Type: Observational
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis
Keywords: psoriasis; microbiota
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control: group of healthy participants
- Topical psoriasis treatment: Group of patients who are treated with topical medications for psoriasis
- Systemic psoriasis treatment: Group of patients who are treated with systematic medications for psoriasis

SUMMARY:
At least 20 psoriasis patients will be compared to at least 20 participants without psoriasis Bacterial genomic DNA will be extracted from stool samples of participants. The intestinal bacterial populations will be compared in order to examine whether there are differences between the groups.

DETAILED DESCRIPTION:
Intestinal bacterial population has a significant influence on health and sickness conditions. It affects the development and the function of the immune system (Th2, Th1 or Th17) by bacterial protein expression and by the composition of the bacterial population.

Psoriasis is an immune related dermal disease. The trigger for this disease is currently unknown but, it is possible that intestinal bacteria are a factor in its development.

Study design:

Participants will be divided into 3 groups:

* Psoriasis patients treated with topical medications
* Psoriasis patients treated with IV or sub-cutaneous medications (e.g biological medications)
* Healthy participants (control group) Bacterial genomic DNA will be extracted from stool samples of participants. The intestinal bacterial populations will be compared in order to examine whether there are differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Dermal psoriasis patients diagnosed by a dermatologist.

Exclusion Criteria:

* Treatment with antibiotics or probiotics within the prior 3 months.
* incapable of signing an inform concent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both psoriasis patients and healthy participants (as a control group) will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
A significant change (P<0.05) in enteric bacterial composition of psoriasis patients (n=20) vs controls (n=20) as assessed by alpha diversity, beta diversity and taxonomic analysis. | 2 years
  To examine whether fecal bacterial populations of psoriasis patients (not treated by enteral medications) are different compared to healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shapiro, Dr., Principal Investigator — Maccabi Healthcare Services, Israel

REFERENCES:
- [Background] Shaw SY, Blanchard JF, Bernstein CN. Association between early childhood otitis media and pediatric inflammatory bowel disease: an exploratory population-based analysis. J Pediatr. 2013 Mar;162(3):510-4. doi: 10.1016/j.jpeds.2012.08.037. Epub 2012 Oct 17. PMID 23084703
- [Background] Shaw SY, Blanchard JF, Bernstein CN. Association between the use of antibiotics in the first year of life and pediatric inflammatory bowel disease. Am J Gastroenterol. 2010 Dec;105(12):2687-92. doi: 10.1038/ajg.2010.398. Epub 2010 Oct 12. PMID 20940708
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131
- [Background] Edgar RC. Search and clustering orders of magnitude faster than BLAST. Bioinformatics. 2010 Oct 1;26(19):2460-1. doi: 10.1093/bioinformatics/btq461. Epub 2010 Aug 12. PMID 20709691
- [Background] Henseler T, Christophers E. Psoriasis of early and late onset: characterization of two types of psoriasis vulgaris. J Am Acad Dermatol. 1985 Sep;13(3):450-6. doi: 10.1016/s0190-9622(85)70188-0. PMID 4056119